CLINICAL TRIAL: NCT01291784
Title: Phase I Study of GC1008 in Patients With Primary Myelofibrosis (PMF), Post-polycythemia Vera/Essential Thrombocythemia Related Myelofibrosis (Post-PV/ET MF)
Brief Title: Anti-TGF-beta Therapy in Patients With Myelofibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Early termination when the drug was no longer made available by the pharmaceutical company due to unanticipated management and administrative decisions.
Sponsor: John Mascarenhas (Other)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 10-1450; GC1008-JM
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Myelofibrosis; Primary Myelofibrosis; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Post-essential Thrombocythemia Related Myelofibrosis
Keywords: monoclonal antibody
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — fresolimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- monoclonal antibody to TGF-beta (Experimental): starting dose of 1mg/kg intravenous over approximately 1 hour every 4 weeks for a total of 6 doses
  Interventions: Biological: monoclonal antibody to TGF-beta

INTERVENTIONS:
Biological: monoclonal antibody to TGF-beta — starting dose of 1mg/kg intravenous over approximately 1 hour every 4 weeks for a total of 6 doses
  Other Names: GC1008

SUMMARY:
TGF-β is a cytokine that is found to be upregulated in the bone marrow of patients with myelofibrosis. This cytokine likely plays a dual role in promoting myelofibrosis and myeloproliferation, both of which are the bone marrow morphologic hallmark of MF. The investigators propose that inhibiting the TGF-β signaling pathway in MF will decrease the fibrogenic stimuli leading to myelofibrosis and concomitantly interrupt myeloproliferation. This is a novel approach to the treatment of patients with myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* ECOG 0-2
* Intermediate-1 or higher by IWG-MRT Post PV/ET MF patients OR intermediate-1 or higher JAK2V617F negative PMF
* Bone marrow MF-2 or higher as assessed by the European consensus grading score AND grade 3 or higher by modified Bauermeister scale.
* Patients must be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney.
* Male and female patients of child-producing potential must agree to use effective contraception while enrolled on study and receiving the investigational agent, and for at least 3 months after the last treatment.
* At the time of enrollment, patients must be >4 weeks since major surgery, radiotherapy, chemotherapy (except hydroxyurea) immunotherapy, or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to < Grade 1, exclusive of alopecia. Concurrent cancer therapy is not permitted for the exception of hydroxyurea if already being used at a stable dose for 3 weeks prior to screening.
* Patients must have negative tests for human immunodeficiency virus (HIV) and for hepatitis viruses B and C (antibody and/or antigen) unless the result is consistent with prior vaccination or prior infection with full recovery.
* Marrow: Absolute neutrophil count ≥ 500/mm3, and platelet count ≥50,000/mm3 without the need for platelet transfusion within 4 weeks
* Hepatic: Serum total bilirubin >1.5 X upper limit of normal (ULN) (Patients with Gilbert's Disease may be included if their total bilirubin is >3.0 mg/dL); alanine aminotransferase (ALT), and aspartate aminotransferase (AST) >2.5 X ULN.
* Renal: Serum creatinine of < 1.5 x upper limit of normal (ULN) or, if higher, estimated or measured creatinine clearance >45 mL/min.
* Coagulation:

  1. Prothrombin Time (PT) < 1.5 X ULN
  2. Partial thromboplastin time (aPTT) < 1.5 X ULN

Exclusion Criteria:

* Central nervous system (CNS) cancer or metastases, meningeal carcinomatosis, malignant seizures, or a disease that either causes or threatens neurologic compromise (e.g., unstable vertebral metastases).
* Pregnant or nursing women, due to the unknown effects of GC1008 on the developing fetus or newborn infant.
* Patients with known bleeding diathesis or signs of uncontrolled active bleeding (hematuria, GI bleeding) other than self-limited causes of benign etiology that have been adequately investigated at the discretion of the investigator.
* Patients requiring anticoagulation with aspirin > 81mg daily, unfractionated heparin, low molecular weight heparin (LMWH), direct anti-thrombin inhibitors, or vitamin K antagonists (e.g. warfarin). This does not apply to patients actively receiving aspirin at a dose of ≤ 81mg a day.
* Patients diagnosed with another malignancy - unless following curative intent therapy, the patient has been disease free for at least 5 years and the probability of recurrence of the prior malignancy is >5%. Patients with curatively treated early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia (CIN) are eligible for this study.
* Patients with an organ transplant, including those that have received an allogeneic bone marrow transplant.
* Use of investigational agents within 4 weeks prior to study enrollment (within 6 weeks if the treatment was with a long-acting agent such as a monoclonal antibody).
* Significant or uncontrolled medical illness, such as congestive heart failure (CHF), myocardial infarction, symptomatic coronary artery disease, significant ventricular arrhythmias within the last 6 months, or significant pulmonary dysfunction. Patients with a remote history of asthma or active mild asthma may participate.
* Active autoimmune disorders or concurrent immunosuppressive medications such as prednisone, interferon, cyclosporine, methotrexate or azathioprine.
* Active infection requiring antibiotics.
* A known allergy to any component of GC1008.
* Patients who, in the opinion of the Investigator, have significant medical or psychosocial problems that warrant exclusion. Examples of significant problems include, but are not limited to:

  1. Other serious non-malignancy-associated medical conditions that may be expected to limit life expectancy or significantly increase the risk of SAEs.
  2. Any condition, psychiatric, substance abuse, or otherwise, that, in the opinion of the Investigator, would preclude informed consent, consistent follow-up, or compliance with any aspect of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Ronald Hoffman, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Mascarenhas J, Li T, Sandy L, Newsom C, Petersen B, Godbold J, Hoffman R. Anti-transforming growth factor-beta therapy in patients with myelofibrosis. Leuk Lymphoma. 2014 Feb;55(2):450-2. doi: 10.3109/10428194.2013.805329. Epub 2013 Jun 24. No abstract available. PMID 23682558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from Jan 2011 to Feb 2012 of known patients to the medical clinic.
Groups:
- Sub A: Subject A
- Sub B: Subject B
- Sub C: Subject C
Period: Overall Study
Arm/Group | Sub A | Sub B | Sub C
Started | 1 | 1 | 1
Completed | 1 | 0 | 1
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: patients with intermediate -1 or higher primary myelofibrosis (PMF) or post-polycythemia vera/essential thrombocythemia myelofibrosis (Post-PV/ET MF). Patients were eligible if they had documented BMF of MF-2 or higher as assessed by the European consensus grading score and grade 3 or higher by modified Bauermeister scale.
Groups:
- Phase 1 MF Subjects: 3 subjects were enrolled in the study. The three subjects were treated at a GC1008 dose level of 1 mg/kg given intravenously over approximately 60 minutes and then repeated every 28 days for a total of 6 cycles in the core study period and then an additional 6 cycles in an extension phase.
Arm/Group | Phase 1 MF Subjects
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Actual age
  years | 68.67 (10.07) [70 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: To assess the safety and tolerability of GC1008 in patients with primary myelofibrosis (PMF) or post-polycythemia vera/essential thrombocythemia myelofibrosis (Post-PV/ET MF).
  A total of 9 AEs determined by the investigator to be at least possibly related to GC1008 occurred during the study.
Time Frame: 28 days
Measure: Number; unit: events
Arm/Group | Sub A | Sub B | Sub C
Number analyzed (Participants) | 1 | 1 | 1
events | 4 | 4 | 1

2. Secondary Outcome: Bauermeister Scale
Description: To assess the clinical response to therapy with GC1008 by International Working Group (IWG) criteria and measure the change in degree of bone marrow fibrosis (BMF) assessed by Bauermeister scale.
  Bauermeister scale: 0, no demonstrable reticulin fibers; 1, occasional fine individual fibers and foci of a fine-fiber network; 2, fine fiber network throughout most of the section, but no coarse fibers; 3, diffuse fiber network with scattered thick coarse fibers, but no mature collagen; and 4, diffuse, often coarse fiber network with areas of collagen.
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | Sub A | Sub B | Sub C
Number analyzed (Participants) | 1 | 1 | 1
units on a scale | 4 | 3 | 4

3. Secondary Outcome: European Consensus Fibrosis Grade
Description: To assess the clinical response to therapy with GC1008 by International Working Group (IWG) criteria and measure the change in degree of bone marrow fibrosis (BMF) assessed by European consensus grading system.
  This scheme consists of a qualitative (reticulin or collagen) and quantitative evaluation of bone marrow fibrosis and distinguishes four increasing categories, ranging from MF-0, which corresponds to normal bone marrow, to MF-3, in which coarse bundles of collagen fibrosis are identifiable with significant osteosclerosis.
Time Frame: 6 months
Measure: Number; unit: units on a scale
Arm/Group | Sub A | Sub B | Sub C
Number analyzed (Participants) | 1 | 1 | 1
units on a scale | 3 | 2 | 2

4. Secondary Outcome: Peripheral Blood CD34+
Description: Investigate exploratory markers for their ability to predict responsiveness to treatment with GC1008.
Time Frame: 6 months
Measure: Number; unit: percentage of hematopoietic stem cells
Arm/Group | Sub A | Sub B | Sub C
Number analyzed (Participants) | 1 | 1 | 1
percentage of hematopoietic stem cells | 3 | 2 | 0

5. Secondary Outcome: JAK2V617F Allele Burden
Description: Investigate exploratory markers, hematopoietic cells, for their ability to predict responsiveness to treatment with GC1008. Analysis of percentage of mutant alleles in hematopoietic stem cells.
Time Frame: 6 months
Measure: Number; unit: percentage of mutant alleles
Arm/Group | Sub A | Sub B | Sub C
Number analyzed (Participants) | 1 | 1 | 1
percentage of mutant alleles | 48 | 95 | 14

ADVERSE EVENTS:
Arm/Group | Sub A | Sub B | Sub C
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub A (N=1) | Sub B (N=1) | Sub C (N=1)
Asystole (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — This event was deemed to not be drug related. Participant progressed to MF
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sub A (N=1) | Sub B (N=1) | Sub C (N=1)
leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
hypoxia (General disorders) | 0 (0) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
skin lesions (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
herpes zoster (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination when the drug was no longer made available by the pharmaceutical company due to unanticipated management and administrative decisions.

Limited patient data (2 evaluable patients), a dose accumulation ratio cannot be determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes